CLINICAL TRIAL: NCT03817099
Title: Effects of Malaysia Diabetes Ramadan Nutrition Plan (My Dia-RNP) on Adherence, Acceptability, Efficacy Potential and Quality of Life in Patients With Type 2 Diabetes Mellitus: A Feasibility Study
Brief Title: Malaysia Diabetes Ramadan Nutrition Plan (My Dia-RNP®): A Feasibility Study
Acronym: MyDia-RNP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Nestle Health Science (Industry); Joslin Diabetes Center (Other)
Responsible Party: Principal Investigator, Barakatun Nisak Bt Mohd Yusof, Associate Professor, Universiti Putra Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MyDia-RNP study
Record Dates: First submitted 2019-01-09; First posted 2019-01-25 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study based on their choice
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- My Dia-RNP (Experimental): In the My Dia-RNP group, participants will undergo the pre-RNP assessment 2 weeks before Ramadan. They will be given a nutrition education based on the Ramadan Nutrition Plan Guide published by IDF-DAR Practical Guidelines. They will also be asked to incorporate diabetes-specific nutrition formula (Nutren untuk Diabetik®) within the prescribed calories before Ramadan period to help them familiarise with a dietary change.
  Interventions: Other: Nutrition Intervention based on My Dia-RNP
- Usual Care (Active Comparator): Participant in this group will continue in a usual care (UC) group. They will receive dietary advice based on the Practical Guide to Diabetes Management in Ramadan produced by Ministry of Health (2015).
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Nutrition Intervention based on My Dia-RNP — Subjects in this group will be advised to follow My Dia-RNP and to incorporate diabetes-specific formula (Nutren®Untuk Diabetik)
  Arms: My Dia-RNP
Other: Usual Care — Subjects in the group continue with the usual care
  Arms: Usual Care

SUMMARY:
Ramadan fasting is an important event for Muslims. During Ramadan, all healthy Muslims are asked to abstain from food and drink throughout the day and eat only during daybreak (also know as Sahur in Malay/Arabic language) and after sunset (also know as Iftar in Malay/Arabic language). Patients with type 2 diabetes (T2DM) can be exempted from fasting but most of them do not perceive themselves as sick, and they continue to fast. With so many Muslims with diabetes choosing to fast, there is an immediate need for evidence-based nutrition practice guidelines. This study is conducted to determine the feasibility of implementing the Ramadan Nutrition Plan named My Dia-RNP that is also incorporating diabetes-specific nutrition formula on dietary adherence and acceptability in patients with type 2 diabetes mellitus. We hypothesized that My Dia-RNP is feasible to be practiced by patients with type 2 diabetes.

DETAILED DESCRIPTION:
In Malaysia, average fasting duration is about 14 hours which could potentially cause hypoglycemia, hyperglycemia, ketoacidosis, and dehydration among people with diabetes. Also, Ramadan triggers a prime dietary change leading to increased risk of nutritional issues from improper eating habits and reduction in physical activity level (Hamdy et al., 2016). Ramadan fasting, therefore, represents a challenge to both patients and healthcare professionals (HCPs) including dietitians.

Ramadan Nutrition Plan (RNP) has recently published by the International Diabetes Federation (IDF) and the Diabetes and Ramadan (DAR) International Alliance IDF-DAR guidelines. The goal is to provide comprehensive guidance on nutrition practice during Ramadan. However, its feasibility in the real clinical scenarios warrants further investigation.

Besides, the use of a diabetes-specific nutrition formula (Nutren Untuk Diabetik®) has been shown beneficial in improving blood glucose control and managing body weight as well as enhancing the nutrient adequacy among people with diabetes (Hamdy and Barakatun-Nisak 2016). While the benefits have been well established, no study has explored its potential during Ramadan.

Malaysia Diabetes-Ramadan Nutrition Plan (My Dia-RNP) is proposed to determine the feasibility of implementing the RNP and to incorporate the diabetes-specific nutrition formula (Nutren Untuk Diabetik®) during Ramadan on dietary adherence and acceptability in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* All Muslim patients aged > 18 years old
* Have a confirmed diagnosis of T2D for at least 6 months
* BMI > 18.5 but < 40 kg/m2
* HbA1c of > 6.5% but < 10%
* On a stabilised dose of oral anti-diabetes agents (OAD) for the past 2 months prior to the study
* Willing to fast for at least 15 days during Ramadan

Exclusion Criteria:

* History of hypoglycaemia leading to hospitalization during the previous Ramadan
* Liver disease
* Abnormal liver function test or renal profiles
* On insulin injection
* Reported abnormal thyroid stimulating hormones
* Use of medications known to effect lipid or glucose metabolism such as steroid
* Pregnancy or the desire to become pregnant in the next 3 months
* On any weight loss program or weight loss medications
* History of cancer undergoing active treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of participants completed the study | 12 weeks
  The ability and likelihood to complete a study successfully with the aim to achieve at least 80% of the study retention rates.

SECONDARY OUTCOMES:
Rate of participants adhered to the intervention | 12 weeks
  Dietary adherence refers to the ability of the participants to adhere to the selected group. This study aims to achieve the completeness of Ramadan Diaries and the able to consume diabetes-specific nutrition formula (Nutren® untuk Diabetik) for at least 75% during the study period.
Efficacy potential on the rate of hypoglycemia | 12 weeks
  Changes in rate of hypoglycemia during Ramadan
Efficacy potential on the fructosamine level | 4 weeks
  Changes in fructosamine levels
Efficacy potential on fasting glucose | 12 weeks
  Changes in fasting blood glucose levels
Efficacy potential on glycemic control | 12 weeks
  Changes in HbA1c levels
Efficacy potential on functional status | 12 weeks
  Changes in hand grip strength
Efficacy potential on body mass index | 12 weeks
  Changes in body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Barakatun-Nisak Mohd Yusof, PhD, Principal Investigator — Universiti Putra Malaysia; Wan Zul Haikal Hafiz Wan Zukiman, Mmed, Principal Investigator — Universiti Putra Malaysia; Noraida Omar, PhD, Principal Investigator — Universiti Putra Malaysia; Zalina Abu Zaid, PhD, Principal Investigator — Universiti Putra Malaysia; Azrina Azlan, PhD, Principal Investigator — Universiti Putra Malaysia; Firdaus Mamat @ Mukhtar, PhD, Principal Investigator — Universiti Putra Malaysia; Norhasmah Sulaiman, PhD, Principal Investigator — Universiti Putra Malaysia; Siti NurA'syura Adznam, PhD, Principal Investigator — Universiti Putra Malaysia; Nur Maziah Hanum Osman, Master, Principal Investigator — Universiti Putra Malaysia; Nor Farahain Yahya, Degree, Principal Investigator — Universiti Putra Malaysia; Osama Hamdy, MD, PhD, Principal Investigator — Joslin Diabetes Centre
Locations (1):
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
The data is subjected to privacy

REFERENCES:
- [Background] Babineaux SM, Toaima D, Boye KS, Zagar A, Tahbaz A, Jabbar A, Hassanein M. Multi-country retrospective observational study of the management and outcomes of patients with Type 2 diabetes during Ramadan in 2010 (CREED). Diabet Med. 2015 Jun;32(6):819-28. doi: 10.1111/dme.12685. Epub 2015 Apr 10. PMID 25581456
- [Background] Bujang MA, Ismail M, Hatta NKBM, Othman SH, Baharum N, Lazim SSM. Validation of the Malay version of Diabetes Quality of Life (DQOL) Questionnaire for Adult Population with Type 2 Diabetes Mellitus. Malays J Med Sci. 2017 Aug;24(4):86-96. doi: 10.21315/mjms2017.24.4.10. Epub 2017 Aug 18. PMID 28951693
- [Background] Campbell M, Fitzpatrick R, Haines A, Kinmonth AL, Sandercock P, Spiegelhalter D, Tyrer P. Framework for design and evaluation of complex interventions to improve health. BMJ. 2000 Sep 16;321(7262):694-6. doi: 10.1136/bmj.321.7262.694. No abstract available. PMID 10987780
- [Background] Hamdy O, Barakatun-Nisak MY. Nutrition in Diabetes. Endocrinol Metab Clin North Am. 2016 Dec;45(4):799-817. doi: 10.1016/j.ecl.2016.06.010. PMID 27823606
- [Background] Lee JY, Wong CP, Tan CSS, Nasir NH, Lee SWH. Type 2 diabetes patient's perspective on Ramadan fasting: a qualitative study. BMJ Open Diabetes Res Care. 2017 May 8;5(1):e000365. doi: 10.1136/bmjdrc-2016-000365. eCollection 2017. PMID 28761651
- [Background] Lee SWH, Lee JY, Tan CSS, Wong CP. Strategies to Make Ramadan Fasting Safer in Type 2 Diabetics: A Systematic Review and Network Meta-analysis of Randomized Controlled Trials and Observational Studies. Medicine (Baltimore). 2016 Jan;95(2):e2457. doi: 10.1097/MD.0000000000002457. PMID 26765440
- [Background] Lee JY, Wong CP, Tan CSS, Nasir NH, Lee SWH. Telemonitoring in fasting individuals with Type 2 Diabetes Mellitus during Ramadan: A prospective, randomised controlled study. Sci Rep. 2017 Aug 31;7(1):10119. doi: 10.1038/s41598-017-10564-y. PMID 28860546
- [Background] Lessan N, Hannoun Z, Hasan H, Barakat MT. Glucose excursions and glycaemic control during Ramadan fasting in diabetic patients: insights from continuous glucose monitoring (CGM). Diabetes Metab. 2015 Feb;41(1):28-36. doi: 10.1016/j.diabet.2014.11.004. Epub 2014 Dec 10. PMID 25497966
- [Background] Salti I, Benard E, Detournay B, Bianchi-Biscay M, Le Brigand C, Voinet C, Jabbar A; EPIDIAR study group. A population-based study of diabetes and its characteristics during the fasting month of Ramadan in 13 countries: results of the epidemiology of diabetes and Ramadan 1422/2001 (EPIDIAR) study. Diabetes Care. 2004 Oct;27(10):2306-11. doi: 10.2337/diacare.27.10.2306. PMID 15451892
- [Background] Hassanein M, Al-Arouj M, Hamdy O, Bebakar WMW, Jabbar A, Al-Madani A, Hanif W, Lessan N, Basit A, Tayeb K, Omar M, Abdallah K, Al Twaim A, Buyukbese MA, El-Sayed AA, Ben-Nakhi A; International Diabetes Federation (IDF), in collaboration with the Diabetes and Ramadan (DAR) International Alliance. Diabetes and Ramadan: Practical guidelines. Diabetes Res Clin Pract. 2017 Apr;126:303-316. doi: 10.1016/j.diabres.2017.03.003. Epub 2017 Mar 12. PMID 28347497
- [Background] Jadviscokova T, Fajkusova Z, Pallayova M, Luza J, Kuzmina G. Occurence of adverse events due to continuous glucose monitoring. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2007 Dec;151(2):263-6. doi: 10.5507/bp.2007.044. PMID 18345261